CLINICAL TRIAL: NCT04449874
Title: A Phase Ia/Ib Dose-Escalation and Dose-Expansion Study Evaluating the Safety, Pharmacokinetics, and Activity of GDC-6036 as a Single Agent and in Combination With Other Anti-cancer Therapies in Patients With Advanced or Metastatic Solid Tumors With a KRAS G12C Mutation
Brief Title: A Study to Evaluate the Safety, Pharmacokinetics, and Activity of GDC-6036 Alone or in Combination in Participants With Advanced or Metastatic Solid Tumors With a KRAS G12C Mutation
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Genentech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: GO42144; 2020-000084-22 (EudraCT Number); 2023-506311-18-00 (Other: EU CT Number)
Record Dates: First submitted 2020-06-24; First posted 2020-06-29 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: Non-Small Cell Lung Cancer; Colorectal Cancer; Advanced Solid Tumors
Keywords: KRAS G12C; Non-Small Cell Lung Cancer; Colorectal Cancer; GDC-6036; Metastatic Solid Tumor; Atezolizumab; Bevacizumab; Cetuximab; Erlotinib; Inavolisib; GDC-1971; SHP2
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Colorectal Neoplasms; Neoplasm Metastasis | interventions — atezolizumab; Cetuximab; Bevacizumab; Erlotinib Hydrochloride; inavolisib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (7):
- Arm A: Dose-escalation (Stage I), Dose Expansion (Stage II) (Experimental): Participants in Stage I will receive GDC-6036 administered orally once daily (PO QD). The dose will be increased in successive cohorts until a study-specific threshold is reached.
  Participants with select solid tumors will be treated with GDC-6036 PO QD in Stage II.
  Interventions: Drug: GDC-6036
- Arm B: GDC-6036 + Atezolizumab (Stage I and Stage II) (Experimental): Participants with non-small cell lung cancer will receive GDC-6036 in combination with atezolizumab.
  Interventions: Drug: GDC-6036; Drug: Atezolizumab
- Arm C: GDC-6036 + Cetuximab (Stage I and Stage II) (Experimental): Participants with colorectal cancer will receive GDC-6036 in combination with cetuximab.
  Interventions: Drug: GDC-6036; Drug: Cetuximab
- Arm D: GDC-6036 + Bevacizumab (Stage I and Stage II) (Experimental): Participants with solid tumors will receive GDC-6036 in combination with bevacizumab.
  Interventions: Drug: GDC-6036; Drug: Bevacizumab
- Arm E: GDC-6036 + Erlotinib (Stage I and Stage II) (Experimental): Participants with non-small cell lung cancer will receive GDC-6036 in combination with erlotinib.
  Interventions: Drug: GDC-6036; Drug: Erlotinib
- Arm F: GDC-6036 + GDC-1971 (Stage I and Stage II) (Experimental): Participants with solid tumors will receive GDC-6036 in combination with GDC-1971 PO in Stage I.
  Participants with select solid tumors will be treated with GDC-6036 in combination with GDC-1971 PO in Stage II.
  Interventions: Drug: GDC-6036; Drug: GDC-1971
- Arm G: GDC-6036 + Inavolisib (Stage I and Stage II) (Experimental): Participants with solid tumors will receive GDC-6036 in combination with inavolisib PO in Stage I.
  Participants with select solid tumors will be treated with GDC-6036 in combination with inavolisib PO in Stage II.
  Interventions: Drug: GDC-6036; Drug: Inavolisib

INTERVENTIONS:
Drug: GDC-6036 — The starting dose of GDC-6036 in the combination Arms B, C, D, E, F and G will be determined from Stage I Arm A (single-agent dose escalation).
Drug: Atezolizumab — A 1200 milligram (mg) intravenous (IV) infusion of atezolizumab will be administered on Day 1 of 21 day cycles.
  Arms: Arm B: GDC-6036 + Atezolizumab (Stage I and Stage II)
Drug: Cetuximab — Cetuximab will be administered at an initial dose of 400 milligram per square meter (mg/m^2) IV infusion followed by 250 mg/m^2 IV infusion weekly in 21 day cycles.
  Arms: Arm C: GDC-6036 + Cetuximab (Stage I and Stage II)
Drug: Bevacizumab — A 15 milligram per kilogram (mg/kg) IV infusion of bevacizumab will be administered on Day 1 of 21 day cycles.
  Arms: Arm D: GDC-6036 + Bevacizumab (Stage I and Stage II)
Drug: Erlotinib — 150 mg of erlotinib will be administered PO QD in 21 day cycles.
  Arms: Arm E: GDC-6036 + Erlotinib (Stage I and Stage II)
Drug: GDC-1971 — The starting dose of GDC-1971 will be determined from its single-agent dose escalation.
  Arms: Arm F: GDC-6036 + GDC-1971 (Stage I and Stage II)
Drug: Inavolisib — The starting dose of inavolisib will be determined from its single-agent dose escalation.
  Arms: Arm G: GDC-6036 + Inavolisib (Stage I and Stage II)

SUMMARY:
This is a Phase I dose-escalation and dose-expansion study that will evaluate the safety, pharmacokinetics (PK), and preliminary activity of GDC-6036 in patients with advanced or metastatic solid tumors with a KRAS G12C mutation.

ELIGIBILITY:
Inclusion Criteria:

* Histologically documented advanced or metastatic solid tumor with KRAS G12C mutation.
* Women of childbearing potential must agree to remain abstinent or use contraception, and agree to refrain from donating eggs during the treatment period and after the final dose of study treatment as specified in the protocol.
* Men who are not surgically sterile must agree to remain abstinent or use a condom, and agreement to refrain from donating sperm during the treatment period and after the final dose of study treatment as specified in the protocol.

Exclusion Criteria:

* Active brain metastases.
* Malabsorption or other condition that interferes with enteral absorption.
* Clinically significant cardiovascular dysfunction or liver disease.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 498 (Estimated)
Dates: Start 2020-07-29 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Percentage of Participants With Adverse Events (AEs) | From Cycle 1 Day 1 until 28 days after the final dose (or as specified in the protocol). A cycle is 21 days.
  Severity is determined according to National Cancer Institute Common Terminology Criteria for Adverse Events, Version 5.0 (NCI CTCAE v5.0)
Percentage of Participants With Dose-Limiting Toxicities (DLTs) | From Cycle 1 Day 1 through Day 21. A cycle is 21 days.

SECONDARY OUTCOMES:
Plasma Concentrations of GDC-6036 | Various timepoints from Cycle 1 Day 1 through study treatment discontinuation (within 28 days after the final dose of study drug). A cycle is 21 days.
Plasma Concentrations of Erlotinib | Various timepoints from Cycle 1 Day 1 through study treatment discontinuation (within 28 days after the final dose of study drug). A cycle is 21 days.
Plasma Concentrations of GDC-1971 | Various timepoints from Cycle 1 Day 1 through study treatment discontinuation (within 28 days after the final dose of study drug). A cycle is 21 days.
Plasma Concentrations of Inavolisib | Various timepoints from Cycle 1 Day 1 through study treatment discontinuation (within 28 days after the final dose of study drug). A cycle is 21 days.
Objective Response Rate (ORR) as Determined by the Investigator According to Response Evaluation Criteria in Solid Tumors, Version 1.1 (RECIST v1.1) | Every 6 weeks from Cycle 1 Day 1 until study treatment discontinuation (within 28 days after the final dose of study drug). A cycle is 21 days.
Duration of Response (DOR) as Determined by the Investigator According to RECIST v1.1 | Every 6 weeks from Cycle 1 Day 1 until study treatment discontinuation (within 28 days after the final dose of study drug). A cycle is 21 days.
Progression-free survival (PFS) as determined by the investigator according to RECIST v1.1 | Every 6 weeks from Cycle 1 Day 1 until study treatment discontinuation (within 28 days after the final dose of study drug). A cycle is 21 days.
Relationship Between GDC-6036 Exposure (Maximum Plasma Concentration Observed [Cmax]) | Various timepoints from Cycle 1 Day 1 through study treatment discontinuation (within 28 days after the final dose of study drug). A cycle is 21 days.
Relationship Between GDC-6036 Exposure (Time to Maximum Plasma Concentration [Tmax]) | Various timepoints from Cycle 1 Day 1 through study treatment discontinuation (within 28 days after the final dose of study drug). A cycle is 21 days.
Relationship Between GDC-6036 Exposure (Half-life [t1/2]) | Various timepoints from Cycle 1 Day 1 through study treatment discontinuation (within 28 days after the final dose of study drug). A cycle is 21 days.
Relationship Between GDC-6036 Exposure (Area Under the Curve [AUC]) | Various timepoints from Cycle 1 Day 1 through study treatment discontinuation (within 28 days after the final dose of study drug). A cycle is 21 days.
Relationship Between Tumor Pharmacodynamic Effects of GDC-6036 | Various timepoints from Cycle 1 Day 1 through study treatment discontinuation (within 28 days after the final dose of study drug). A cycle is 21 days.

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Genentech, Inc.
Locations (63):
- United States (8):
  - City of Hope Comprehensive Cancer Center, Duarte, California
  - UCSD Moores Cancer Center, La Jolla, California
  - Chao Family Comprehensive Cancer Center UCI, Orange, California
  - Yale Cancer Center, New Haven, Connecticut
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - University of Oklahoma, Oklahoma City, Oklahoma
  - Abramson Cancer Center, Philadelphia, Pennsylvania
  - UPMC - Hillman Cancer Center, Pittsburgh, Pennsylvania
- Australia (5):
  - St Vincent's Hospital Sydney, Darlinghurst, New South Wales
  - Slade Health Inward goods, Mount Kuring-Gai, New South Wales
  - Peter MacCallum Cancer Center, Melbourne, Victoria
  - Alfred Health, Melbourne, Victoria
  - Linear Clinical Research Limited, Nedlands, Western Australia
- Belgium (3):
  - UZ Antwerpen, Edegem
  - CHU de Liège, Liège
  - AZ St Maarten Campus Leopoldstr, Mechelen
- Brazil (6):
  - Santa Casa de Misericordia de Belo Horizonte - PPDS, Belo Horizonte, Minas Gerais
  - Hospital Erasto Gaertner, Curitiba, Paraná
  - Hospital de Clinicas de Porto Alegre HCPA PPDS, Pôrto Alegre, Pará
  - Universidade de Caxias do Sul, Caxias do Sul, Rio Grande do Sul
  - Hospital Sao Lucas Da Pontificia Universidade Catolica Do Rio Grande Do Sul (PUCRS), Porto Alegre, Rio Grande do Sul
  - Instituto Nacional de Câncer, Rio de Janeiro
- Canada (3):
  - Ottawa Hospital, Ottawa, Ontario
  - Princess Margaret Cancer Centre, Toronto, Ontario
  - Jewish General Hospital, Montreal, Quebec
- Clinexpert Gyongyos Kft, Gyöngyös, Hungary
- Israel (3):
  - Rambam Medical Center, Haifa
  - Sheba Medical Center - PPDS, Ramat Gan
  - Tel-Aviv Sourasky Medical Center, Tel Aviv
- Italy (5):
  - Istituto Scientifico Romagnolo Per Lo Studio E La Cura Dei Tumori IRST - PPDS, Meldola, Emilia-Romagna
  - Irccs Ospedale San Raffaele, Milan, Lombardy
  - Asst Grande Ospedale Metropolitano Niguarda, Milan, Lombardy
  - Istituto Clinico Humanitas, Rozzano (MI), Lombardy
  - Azienda Ospedaliero Universitaria Pisana, Pisa, Tuscany
- The Aga Khan University-Kenya., Nairobi, Kenya
- Netherlands (4):
  - Het Nederlands Kanker Instituut Antoni Van Leeuwenhoek Ziekenhuis, Amsterdam
  - Leids Universitair Medisch Centrum, Leiden
  - Maastricht University Medical Center, Maastricht
  - Universitair Medisch Centrum Utrecht, Utrecht
- New Zealand (3):
  - Auckland City Hospital, Cancer and Blood Research, Auckland
  - Auckland City Hospital, Auckland
  - New Zealand Clinical Research - Christchurch, Christchurch
- Norway (2):
  - Haukeland University Hospital, Bergen
  - Oslo university hospital Radiumhospitalet, Oslo
- Poland (2):
  - Uniwersyteckie Centrum Kliniczne, O?rodek Bada? Klinicznych Wczesnych Faz, Gdansk
  - Biokinetica, Przychodnia Jozefow, Józefów
- South Korea (4):
  - Seoul National University Bundang Hospital, Seongnam-si
  - Seoul National University Hospital, Seoul
  - Asan Medical Center - PPDS, Seoul
  - Samsung Medical Center - PPDS, Seoul
- Spain (7):
  - Hospital Universitari Vall d'Hebron, Barcelona
  - START Madrid-FJD, Hospital Fundacion Jimenez Diaz, Madrid
  - Hospital Universitario 12 de Octubre, Madrid
  - Hospital Universitario HM Sanchinarro-CIOCC, Madrid
  - Hospital Clinico Universitario Virgen de la Victoria, Málaga
  - Hospital Universitario Virgen del Rocío, Seville
  - Hospital Clinico Universitario de Valencia, Valencia
- Switzerland (2):
  - Inselspital, Bern
  - Hôpitaux Universitaires de Genève, Geneva
- United Kingdom (4):
  - Queen Elizabeth Hospital, Birmingham
  - Velindre Cancer Centre, Cardiff
  - University College London Hospitals NHS Foundation Trust, London
  - The Christie NHS Foundation Trust, Manchester

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Sacher AG, Miller WH Jr, Patel MR, Paz-Ares L, Santoro A, Ahn MJ, Dziadziuszko R, Freres P, Luo J, Bowyer S, Desai J, Markman B, De Miguel M, Deva S, Falcon A, Alonso G, Guedes JD, Kim SH, Krebs MG, Laurie SA, Massarelli E, Medina L, Prenen H, Amatu A, Van Dongen M, Choi Y, Hou X, Qi T, Lin MT, Koli K, Mayo MC, Yau KK, Royer-Joo S, Chang J, Jun T, Dharia NV, Schutzman JL, Lorusso P; GO42144 Investigator Study group; GO42144 Investigator Study Group. Single-Agent Divarasib in Patients With KRAS G12C-Positive Non-Small Cell Lung Cancer: Long-Term Follow-Up of a Phase I Study. J Clin Oncol. 2025 Oct 20;43(30):3249-3253. doi: 10.1200/JCO-25-00040. Epub 2025 Jul 9. PMID 40632992
- [Derived] Desai J, Alonso G, Kim SH, Cervantes A, Karasic T, Medina L, Shacham-Shmueli E, Cosman R, Falcon A, Gort E, Guren T, Massarelli E, Miller WH Jr, Paz-Ares L, Prenen H, Amatu A, Cremolini C, Kim TW, Moreno V, Ou SI, Passardi A, Sacher A, Santoro A, Stec R, Ulahannan S, Arbour K, Lorusso P, Luo J, Patel MR, Choi Y, Shi Z, Mandlekar S, Lin MT, Royer-Joo S, Chang J, Jun T, Dharia NV, Schutzman JL; GO42144 Investigator and Study Group; Han SW. Divarasib plus cetuximab in KRAS G12C-positive colorectal cancer: a phase 1b trial. Nat Med. 2024 Jan;30(1):271-278. doi: 10.1038/s41591-023-02696-8. Epub 2023 Dec 5. PMID 38052910
- [Derived] Sacher A, LoRusso P, Patel MR, Miller WH Jr, Garralda E, Forster MD, Santoro A, Falcon A, Kim TW, Paz-Ares L, Bowyer S, de Miguel M, Han SW, Krebs MG, Lee JS, Cheng ML, Arbour K, Massarelli E, Choi Y, Shi Z, Mandlekar S, Lin MT, Royer-Joo S, Chang J, Dharia NV, Schutzman JL, Desai J; GO42144 Investigator and Study Group. Single-Agent Divarasib (GDC-6036) in Solid Tumors with a KRAS G12C Mutation. N Engl J Med. 2023 Aug 24;389(8):710-721. doi: 10.1056/NEJMoa2303810. PMID 37611121